CLINICAL TRIAL: NCT05846711
Title: The Accuracy of Manual BPPV Diagnostics: A Randomized Crossover Study With Comparison of Manual Diagnostic and Diagnostic in TRV Chair, When Using VNG Goggles in Both Scenarios.
Brief Title: The Accuracy of Manual BPPV Diagnostics When Using VNG Goggles.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Malene Hentze Hansen, Principal Investigator, Aalborg University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 20220061
Record Dates: First submitted 2023-04-17; First posted 2023-05-06 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Benign Paroxysmal Positional Vertigo; BPPV; Vertigo; Vestibular Disorder; Vestibular Diseases; Labyrinth Diseases; Inner Ear Disease
Keywords: TRV reposition chair; Dix-Hallpike maneuver; Supine Roll Test
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Vestibular Diseases; Labyrinth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bedside BPPV diagnostics (Active Comparator): Diagnostics of BPPV with manual tests using VNG goggles. The goggles will be added an IMU sensor detecting angulation and velocity (the physician will not get feedback from the sensor during the examination. This will only be used in later analysis).
  Interventions: Diagnostic Test: BPPV diagnostic; Device: VNG goggles; Device: IMU sensor; Procedure: Manual BPPV diagnostics
- TRV BPPV diagnostics (Active Comparator): Diagnostics of BPPV using the TRV chair.
  Interventions: Diagnostic Test: BPPV diagnostic; Device: TRV chair; Device: VNG goggles

INTERVENTIONS:
Diagnostic Test: BPPV diagnostic — Supine Roll Test and Dix-Hallpike Test
Device: TRV chair — Mechanical rotational chair
  Arms: TRV BPPV diagnostics
Device: VNG goggles — Goggles for video nystagmography
Device: IMU sensor — A sensor that measures triaxial acceleration and triaxial angular velocity.
  Arms: Bedside BPPV diagnostics
Procedure: Manual BPPV diagnostics — Bedside BPPV diagnostics
  Arms: Bedside BPPV diagnostics

SUMMARY:
The aim is to investigate the accuracy of manual diagnostics of benign paroxysmal positional vertigo (BPPV) by comparing it to BPPV diagnostics in mechanical rotational chair (TRV chair). VNG (videonystagmography) goggles will be used in both scenarios.

Furthermore, the investigators will examine the importance of angulation and velocity in relation to the diagnostic outcome.

DETAILED DESCRIPTION:
Open-label, randomized controlled trial with cross over comparing manual bedside BPPV diagnostics with diagnostics in a mechanical rotational chair (TRV chair) when using VNG goggles in both scenarios.

Patients with a history of positional vertigo will be considered for enrollment and randomized to which diagnostic modality they begin with. Each subject will wait for minimum 30 minutes between the two diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Classic BPPV-patient history (short lasting (<1 minute) positional rotatory vertigo, no accompanying tinnitus or hearing loss, and no focal neurological findings.
* Understand written and spoken Danish

Exclusion Criteria:

* Pregnancy
* Weight ≥ 150 kg and or Height ≥ 2m
* Neck and spine immobility to a degree where MD on examination bed is impossible
* Insufficient cooperation during diagnostic testing
* Sedative antihistamines taken within the past seven days
* Comorbidities: Heart failure (EF < 40), known cerebral aneurysm, cerebrovascular events (<3 months) or dissection disease
* Spontaneous or gaze evoked nystagmus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy | 2 year
  Sensitivity, specificity, positive predictive value and negative predictive value of bedside examination (index-test). Gold standard is diagnostics in the TRV chair.

SECONDARY OUTCOMES:
Head angulation during diagnostic bedside examination. | 2 year
  Angulation of the head during diagnostic bedside examination will be measured using an IMU sensor. Data will be presented as the difference in head angulation compared to the ideal angulation descriped for the diagnostic tests.
Angular velocity during diagnostic bedside examination | 2 year
  Angular velocity of the head movements during diagnostic bedside examination will be measured using an IMU sensor. Data will be presented as mean velocity and peak velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Malene Hentze Hansen, MD, Principal Investigator — Department of Otolaryngology, Head & Neck Surgery and Audiology
Locations (1):
- Department of Otolaryngology, Head & Neck Surgery and Audiology, Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hentze M, Hougaard DD, Kingma H. Impact of head orientation and head movement in traditional manual diagnostics of benign paroxysmal positional vertigo: a randomized controlled crossover study. Front Neurol. 2025 Oct 3;16:1654404. doi: 10.3389/fneur.2025.1654404. eCollection 2025. PMID 41111959
- [Derived] Hentze M, Hougaard DD, Kingma H. The Intra-Examiner Variability in and Accuracy of Traditional Manual Diagnostics of Benign Paroxysmal Positional Vertigo: A Prospective Observational Cohort Study. J Clin Med. 2025 Jan 11;14(2):434. doi: 10.3390/jcm14020434. PMID 39860440
- [Derived] Hentze M, Hougaard DD, Kingma H. Is diagnostics of Benign Paroxysmal Positional Vertigo with a mechanical rotation chair superior to traditional manual diagnostics? A randomized controlled crossover study. Front Neurol. 2024 Dec 6;15:1519837. doi: 10.3389/fneur.2024.1519837. eCollection 2024. PMID 39711790